CLINICAL TRIAL: NCT01240785
Title: Metformin Versus Insulin in Gestational Diabetes. A Randomized Controlled Single Center Trial.
Brief Title: Metformin Versus Insulin in Gestational Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tapani Rönnemaa, professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 246/2005
Record Dates: First submitted 2010-11-03; First posted 2010-11-15 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; metformin; insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Metformin; Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): Metformin 500 mg 1-2 tablets twice daily according to plasma glucose values
  Interventions: Drug: metformin
- insulin (Active Comparator): NPH insulin once or twice daily and/or insulin lispro or aspart according to preprandial and postprandial glucose values
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: metformin — metformin 1 g twice daily or maximum tolerated dose less than 2 g daily
  Other Names: Diformin retard 500 mg
  Arms: Metformin
Drug: insulin — subcutaneous Neutral Protamine Hagedorn (NPH) insulin and/or rapid acting insulin analog adjusted according to plasma glucose values until delivery
  Other Names: Protaphane; Humalog
  Arms: insulin

SUMMARY:
Gestational diabetes is traditionally treated with insulin. Metformin is a peroral drug used worldwide in the treatment of type 2 diabetes and also in a few studies on patients with gestational diabetes. The investigators aim is to compare insulin and metformin in the treatment of gestational diabetes. The investigators hypothesis is that there is no difference between insulin and metformin treated mothers in the main outcome criteria (birth weight, neonatal complications).

DETAILED DESCRIPTION:
Gestational diabetes is traditionally treated with insulin. Metformin is a peroral drug used worldwide in the treatment of type 2 diabetes and also in a few studies on patients with gestational diabetes. The investigators aim is to compare insulin and metformin in the treatment of gestational diabetes. The investigators hypothesis is that there is no difference between insulin and metformin treated mothers in the main outcome criteria (birth weight, neonatal complications). The study was performed as a randomized controlled trial in one center, Turku University hospital using the non-inferiority design in June 2006 - December 2010. The final study population consisted of altogether 217 women, of whom 110 received metformin and 107 insulin.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with gestational diabetes who had at least twice plasma glucose at fasting > 5.4 mmol/L and/or 1 hour postprandial value > 7.7 mmol/L at 24 to 32 gestational weeks

Exclusion Criteria:

1. Fasting glucose > 7.0 mmol/L or 1 hour postprandial plasma glucose > 11.0 mmol/L or Glycosylated hemoglobin A1c (HbA1c) > 7.0%
2. Renal, hepatic or cardiac failure
3. Pregestational use of metformin
4. Pregnancy with multiple fetuses

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2006-06; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapani Rönnemaa, MD, PhD, Principal Investigator — Professor, Chief Physician

REFERENCES:
- [Derived] Huhtala MS, Ronnemaa T, Pellonpera O, Tertti K. Cord serum metabolome and birth weight in patients with gestational diabetes treated with metformin, insulin, or diet alone. BMJ Open Diabetes Res Care. 2021 May;9(1):e002022. doi: 10.1136/bmjdrc-2020-002022. PMID 34059525
- [Derived] Huhtala MS, Tertti K, Juhila J, Sorsa T, Ronnemaa T. Metformin and insulin treatment of gestational diabetes: effects on inflammatory markers and IGF-binding protein-1 - secondary analysis of a randomized controlled trial. BMC Pregnancy Childbirth. 2020 Jul 11;20(1):401. doi: 10.1186/s12884-020-03077-6. PMID 32652973
- [Derived] Huhtala MS, Tertti K, Pellonpera O, Ronnemaa T. Amino acid profile in women with gestational diabetes mellitus treated with metformin or insulin. Diabetes Res Clin Pract. 2018 Dec;146:8-17. doi: 10.1016/j.diabres.2018.09.014. Epub 2018 Sep 15. PMID 30227169
- [Derived] Pellonpera O, Ronnemaa T, Ekblad U, Vahlberg T, Tertti K. The effects of metformin treatment of gestational diabetes on maternal weight and glucose tolerance postpartum--a prospective follow-up study. Acta Obstet Gynecol Scand. 2016 Jan;95(1):79-87. doi: 10.1111/aogs.12788. Epub 2015 Nov 8. PMID 26439816
- [Derived] Tertti K, Laine K, Ekblad U, Rinne V, Ronnemaa T. The degree of fetal metformin exposure does not influence fetal outcome in gestational diabetes mellitus. Acta Diabetol. 2014 Oct;51(5):731-8. doi: 10.1007/s00592-014-0570-6. Epub 2014 Mar 16. PMID 24633859

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin Arm | Insulin
Started | 111 | 110
Completed | 110 (110 women completed in the metformin arm and 107 women completed in the insulin arm.) | 107
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Insulin | Total
Number analyzed (Participants) | 110 | 107 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (5.0) | 32.1 (5.4) | 32.0 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 107 | 217
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 110 | 107 | 217

OUTCOME MEASURES:

1. Primary Outcome: Birth Weight Per Arm
Description: birth weight adjusted for gestational weeks expressed as standard deviation units using data from Finnish fetal growth charts in normal pregnancies
Time Frame: delivery
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
g | 3604 (488) | 3589 (448)

2. Secondary Outcome: Pregnancy Induced Hypertension Per Arm
Description: Participants with pregnancy induced hypertension defined as blood pressure over 140/90 mmHg or increase in systolic blood pressure > 30 mmHg or diastolic blood pressure > 15 mmHg
Time Frame: up to on the average 40 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
participants | 2 | 4

3. Secondary Outcome: Maternal Weight Gain Per Arm
Time Frame: up to on the average 40 weeks of gestation
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
kg | 8.0 (5.3) | 7.9 (5.3)

4. Secondary Outcome: Pre-eclampsia Per Arm
Time Frame: up to on the average 40 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
participants | 5 | 10

5. Secondary Outcome: Mode of Delivery Per Arm
Time Frame: delivery
Measure: Number; unit: no of cesarean section
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
no of cesarean section | 15 | 18

6. Secondary Outcome: Gestational Weeks at Delivery Per Arm
Time Frame: delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
weeks | 39.2 (1.4) | 39.3 (1.6)

7. Secondary Outcome: Induction of Delivery Per Arm
Time Frame: delivery
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
participants | 42 | 58

8. Secondary Outcome: Shoulder Dystocia Per Arm
Time Frame: delivery
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 110 | 107
participants | 1 | 2

9. Secondary Outcome: Neonatal Hypoglycemia Per Arm
Time Frame: 0-24 h after delivery
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 109 | 107
participants | 18 | 18

10. Secondary Outcome: Neonatal Hyperbilirubinemia Per Arm
Time Frame: 0-3 days after delivery
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 109 | 107
participants | 9 | 10

11. Secondary Outcome: Apgar Score at 5 Min After Delivery Per Arm
Description: Apgar score 0-10. 0-2 points from heart rate; 0-2 points for respiratory effort; 0-2 points for skin colour; 0-2 points for muscle tone; 0-2 points for reflex response. For all items the higher the value, the better the outcome
Time Frame: 5 minutes after delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 109 | 107
units on a scale | 8.7 (1.3) | 8.9 (1.0)

12. Secondary Outcome: Neonate Transfer to Intensive Care Unit Per Arm
Time Frame: 0-5 days after delivery
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 109 | 107
participants | 34 | 39

13. Secondary Outcome: Child Outcome at 2 Years Per Arm
Description: neuropsychological and motor skills testing
Time Frame: 2 years after birth
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Fetal cardiac function evaluated with ultrasound and cardiotokography
Arm/Group | Metformin | Insulin
Serious Adverse Events (participants affected / at risk) | 1/110 | 0/107
Other Adverse Events (participants affected / at risk) | 0/110 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=110) | Insulin (N=107)
fetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Fetal death at 39 weeks due to umbilical cord complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No